CLINICAL TRIAL: NCT02082769
Title: A Phase 3, Randomized, Multicenter, Allopurinol-Controlled Study Assessing the Safety and Efficacy of Oral Febuxostat in Subjects With Gout
Brief Title: Safety and Efficacy of Oral Febuxostat in Subjects With Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Qingdao Shengbang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFDA2010L04287
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-03

CONDITIONS: Gout
Keywords: Gout; Uric Acid; Xanthine oxidase; Febuxostat
MeSH Terms: conditions — Gout | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Febuxostat 40 mg QD (Experimental): Febuxostat 40 mg, orally, once daily for up to 24 weeks
  Interventions: Drug: Febuxostat
- Febuxostat 80 mg QD (Experimental): Febuxostat 80 mg, orally, once daily for up to 24 weeks
  Interventions: Drug: Febuxostat
- Allopurinol 100mg QD (Active Comparator): Allopurinol 100mg, orally, three times daily for up to 24 weeks
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat
  Arms: Febuxostat 40 mg QD; Febuxostat 80 mg QD
Drug: Allopurinol
  Arms: Allopurinol 100mg QD

SUMMARY:
The purpose of this study is to compare febuxostat allopurinol in subjects with gout.

DETAILED DESCRIPTION:
A randomized, double-blind, multicenter, allopurinol-controlled and parallel-assigned study comparing 40 mg, 80 mg of febuxostat, and allopurinol 300 mg in subjects with gout. Subjects will receive treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemia (serum urate ≥8.0 mg/dL) and gout by Chinese Rheumatism Association Criteria;
* Renal function defined as a serum creatinine level of < 2.0 mg/dL and creatinine clearance of > 20 milliliters per minute (mL/min) by Cockcroft and Gault formula;
* No gout flare 2 weeks beforehand during 2-week screening period.

Exclusion Criteria:

* Pregnancy or lactation;
* Concurrent therapy with urate lowering agents, azathioprine, 6-mercaptopurine, thiazide diuretics, or medications containing aspirin (>325 mg) or other salicylates;
* Body Mass Index (BMI) >50 kilogram per meter²(kg/m²);
* A history of active liver disease, or hepatic dysfunction;
* A history of bronchial asthma;
* A history of renal calculi or thyroid disease;
* Secondary gout Joint diseases induced by rheumatoid arthritis, psoriatic arthritis and bone tumor;
* Intolerance to allopurinol and Ibuprofen;
* Alcohol intake of ≥ 14 drinks/week;
* Clinically significant medical condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shenren Chen, M.D., Principal Investigator — Second Affiliated Hospital of Shantou University Medical College; Yangang Wang, M.D., Principal Investigator — The Affiliated Hospital of Qingdao University; Xiumei Liu, M.D., Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Hong Liu, M.D., Principal Investigator — First Affiliated Hospital of Guangxi Medical University; Yongde Peng, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Jianqin Wang, M.D., Principal Investigator — Lanzhou University Second Hospital; Jinying Lin, M.D., Principal Investigator — People's Hospital of Guangxi Zhuang Autonomous Region; Haiwang Ji, M.D., Principal Investigator — Shaanxi Provincial People's Hospital; Bin Liu, M.D., Principal Investigator — The First Hospital of Jilin University; Ying Lu, M.D., Principal Investigator — Zhejiang Provincial Tongde Hospital; Peng Liu, M.D., Principal Investigator — Guangxi Ruikang Hospital; Yonghong Zhang, M.D., Principal Investigator — Luoyang Orthopedic-Traumatological Hospital

REFERENCES:
- [Derived] Xu S, Liu X, Ming J, Chen S, Wang Y, Liu X, Liu H, Peng Y, Wang J, Lin J, Ji H, Liu B, Lu Y, Liu P, Zhang Y, Ji Q. A phase 3, multicenter, randomized, allopurinol-controlled study assessing the safety and efficacy of oral febuxostat in Chinese gout patients with hyperuricemia. Int J Rheum Dis. 2015 Jul;18(6):669-78. doi: 10.1111/1756-185X.12648. Epub 2015 May 27. PMID 26013187

RESULTS

PARTICIPANT FLOW:
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg, orally, once daily for up to 24 weeks
  Febuxostat
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily for up to 24 weeks
  Febuxostat
- Allopurinol 100mg QD: Allopurinol 100mg, orally, three times daily for up to 24 weeks
  Allopurinol
Period: Overall Study
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD
Started | 168 | 168 | 168
Completed | 144 | 141 | 132
Not Completed | 24 | 27 | 36

BASELINE CHARACTERISTICS:
Population: full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD | Total
Number analyzed (Participants) | 160 | 158 | 159 | 477
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 160 | 158 | 159 | 477
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.9) | 48.2 (12.0) | 46.5 (10.7) | 46.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 146 | 149 | 453
  Male | 2 | 12 | 10 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (2.7) | 25.1 (2.6) | 25.4 (3.3) | 25.2 (2.8)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 126.2 (10.0) | 126.4 (11.0) | 124.8 (10.1) | 126.4 (10.4)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 79.1 (8.2) | 77.6 (8.1) | 78.7 (7.9) | 78.5 (8.1)
Baseline serum urate level units [Mean (Standard Deviation); unit: umol/l] | 560.8 (73.3) | 565.1 (75.5) | 574.2 (77.8) | 566.7 (75.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Last Three Serum Urate Levels Are <6.0 Milligram Per Deciliter (mg/dL)
Time Frame: Last 3 visits (any last 3 visits up to week 26)
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD
Number analyzed (Participants) | 160 | 158 | 159
percentage of participants | 22.5 | 33.5 | 17.0

2. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Final Visit
Time Frame: Final Visit (up to 26 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD
Number analyzed (Participants) | 160 | 158 | 159
percentage of participants | 45.0 | 58.9 | 34.6

3. Other Pre Specified Outcome: Absolute Change in the Serum Urate Level at the Final Visit Relative to Baseline
Time Frame: Baseline and Final Visit (up to 26 weeks)
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD
Number analyzed (Participants) | 160 | 158 | 159
umol/l | 182.2 (115.6) | 216.0 (137.2) | 170.4 (132.6)

ADVERSE EVENTS:
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Allopurinol 100mg QD
Serious Adverse Events (participants affected / at risk) | 0/168 | 1/168 | 0/168
Other Adverse Events (participants affected / at risk) | 45/168 | 46/168 | 41/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat 40 mg QD (N=168) | Febuxostat 80 mg QD (N=168) | Allopurinol 100mg QD (N=168)
hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — The subject was diagnosed as hydronephrosis after 14-day period of febuxostat administration and thus hospitalized.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat 40 mg QD (N=168) | Febuxostat 80 mg QD (N=168) | Allopurinol 100mg QD (N=168)
Liver function test abnormalities (Hepatobiliary disorders) | 17 (17) | 22 (22) | 18 (18)
Renal function test abnormalities (Renal and urinary disorders) | 2 (2) | 7 (7) | 2 (2)
Abnormal electrocardiogram (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Abnormal urine protein (Renal and urinary disorders) | 4 (4) | 4 (4) | 1 (1)
Drug allergy (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 5 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Others (General disorders) | 12 (12) | 10 (10) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No